CLINICAL TRIAL: NCT02122016
Title: Weaning With Smartcare in Mechanically Ventilated Patients in the ICU - a Controlled and Randomized Study
Brief Title: Comparison of Two Different Types of Mechanical Ventilation Weaning in Patients in the ICU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Corinne Taniguchi, Physiotherapist, PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SmartCare\HIAE11
Record Dates: First submitted 2013-08-27; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Weaning Failure
Keywords: Ventilator weaning; Protocols; Computer driven weaning; Decision Making, Computer-Assisted; Therapy, Computer-Assisted; Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SmartCare (Experimental): A computer driven weaning ventilator, using closed-loop ventilation, taking into account patients lung mechanics and exhaled CO2.
  Interventions: Device: SmartCare
- Conventional weaning protocol (Active Comparator): A conventional weaning protocol consisting of a daily weaning screen, which is performed by physiotherapist. All patients who are mechanically ventilated for more than 24 hours are given a spontaneous breathing trial.
  Interventions: Other: Conventional weaning protocol

INTERVENTIONS:
Device: SmartCare — Ventilator with a SmartCare module that is capable of performing a computer-driven weaning trial taking into account patients lung mechanics and exaled CO2.
  Arms: SmartCare
Other: Conventional weaning protocol — A conventional weaning protocol performed by physiotherapist with a daily weaning screen and a spontaneous breathing trial
  Arms: Conventional weaning protocol

SUMMARY:
Mechanical ventilation is widely used for ICU patients as a lifesaving procedure. However, it is associated with several complications, such as ventilator-associated pneumonia and the increase of hospital morbidity and mortality. To avoid such complications, we need to wean these patients off the ventilator as soon as possible. This must however be done at the right time to avoid other complications, such as the need for re-intubation. For this reason, it is important to have a specific weaning protocol, which will reduce the time on mechanical ventilation, and avoiding the need for re-intubation and other complications. Recently, an argument has developed as to which weaning protocol would be more appropriated, and whether a computer driven weaning protocol could have better results than the conventional weaning protocols focusing on daily screening and daily interruption of sedation followed by a spontaneous breathing test. Our objective is to compare mechanical ventilation times, weaning success up to 48 hours after extubation, re-intubation rates between a group with computer driven weaning protocol (SmartCare) versus a weaning protocol with daily weaning screens and spontaneous breathing trials in ICU patients ventilated for more than 24 hours.

DETAILED DESCRIPTION:
Background: Mechanical ventilation (MV) weaning is commonly performed using Spontaneous Breathing Trials (SBT) with pressure support ventilation after a daily weaning screen [1]. Recently there has been an increased interest in automatic weaning trials, which consists of closed-loop ventilation, using ETCO2 monitoring during SBT [1, 2]. So far, there has been no clinical evidence to compare automatic weaning trials with those of SBT.

Objective: To compare MV weaning times between an Automatic Weaning Ventilation System (SmartCare/PS) and SBT groups.

Methods: A randomized, controlled study performed at a general ICU. Adult patients were enrolled who were ventilated for more than 24 hours. Tracheostomies patients, those with neurological conditions, and a Glasgow coma scales lower than 10 were excluded. Patients were randomized to either the control or Smart Care group. All patients were ventilated with a Drager Evita XL (Drager Medical, Lubeck, Germany) ventilator with SmartCare/PS software version 1.1 available for use immediately prior to randomization. The Control group consisted of a daily weaning screen and SBT with pressure support ventilation. If patients tolerated SBT, they were extubated. Smart Care group patients were also submitted to a daily weaning screen, after which they were ventilated with the SmartCare/PS mode. MV and weaning time, maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP), vital capacity (VC), respiratory frequency to tidal volume ration (f/Vt), use of non-invasive ventilation (NIV) post extubation, and re-intubation rate we evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Recovery from the causes that had led to mechanical ventilation
* Capacity to initiate a spontaneous breathing effort
* Spontaneous eye opening and responsiveness even with low doses of sedation
* Oxygen inspired fraction lower than 50% with oxygen pulse oximeter higher than 95%
* Positive end-expiratory pressure under 10 cmH2O
* Hemodynamic stability
* Vasopressor drugs lower than 0.05mcg/ml/kg

Exclusion Criteria:

* Tracheotomized patients
* Neurological sequels with a poor prognostic (post cardiorespiratory arrest or central neurological injury)
* Glasgow scale lower than 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Weaning time from mechanical ventilation | From June 2011 to April 2012 an 11 month period
  The duration that patient's received mechanical ventilation until they were extubated comparing two weaning protocols (computer driven v daily weaning screen and spontaneous breathing trial).

SECONDARY OUTCOMES:
weaning success | From June 2011 to April 2012 an 11 month period
  Evaluate the rate of weaning success of patients under mechanical ventilation. Success defined as patient not needing re-intubation up to 48 hours after extubation.
re-intubation rate | From June 2011 to April 2012 an 11 month period
  Evaluate the re-intubation rate of patients that were extubated.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Taniguchi, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (2):
- Brazil (2):
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein's Critically Ill Department, São Paulo, São Paulo

REFERENCES:
- [Derived] Taniguchi C, Victor ES, Pieri T, Henn R, Santana C, Giovanetti E, Saghabi C, Timenetsky K, Caserta Eid R, Silva E, Matos GF, Schettino GP, Barbas CS. Smart Care versus respiratory physiotherapy-driven manual weaning for critically ill adult patients: a randomized controlled trial. Crit Care. 2015 Jun 11;19(1):246. doi: 10.1186/s13054-015-0978-6. PMID 26580673